CLINICAL TRIAL: NCT06786936
Title: Evaluating the Role of IL-17 as an Orchestrator of Peripheral-central Cross Talk in Depressive Symptoms
Acronym: ELATE
Status: Recruiting | Type: Observational
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other); Medical Research Council (Other Government)
Responsible Party: Sponsor
Other Study IDs: GN22MH376
Record Dates: First submitted 2025-01-09; First posted 2025-01-22 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Psoriatic Arthritis; Depression; Psoriatic Plaque
MeSH Terms: conditions — Arthritis, Psoriatic; Depression | interventions — secukinumab; bimekizumab; ixekizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be used for peripheral immunophenotyping. This will include the capacity for future proteomic analysis, transcriptomic analysis, epigenetic analysis and flow cytometry.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Psoriatic Disease: Encompasses both Psoriatic Arthritis and and Plague Psoriasis .
  Interventions: Drug: Secukinumab; Drug: Bimekizumab; Drug: Ixekizumab; Drug: Placebo

INTERVENTIONS:
Drug: Secukinumab — Initial dosing of Secukinimab at week 0, 1, 2, 3, 4 and maintenance doses will be determined by the standard care team. This will be 150mg or 300mg. This will be administered by the study team once confirmed and randomisation has occurred for secukinimab/ placebo allocation.
  Other Names: N/A (Not applicable)
Drug: Bimekizumab — Initial dosing of bimkizumab at week 0 & 4 and maintenance doses will be determined by the standard care team. This will be 160mg or 320mg. This will be administered by the study team once confirmed and randomisation has occurred for bimekizumab/ placebo allocation.
  Other Names: N/A (Not applicable)
Drug: Ixekizumab — Initial dosing of Ixekizumab at week 0 & 4 or week 0, 2 & 4, maintenance doses will be determined by the standard care team. The initial dose will be 160mgs then 80mg dose will either be given 2 or 4 weekly. This will be administered by the study team once confirmed and randomisation has occurred for Ixekizumab/ placebo allocation.
  Other Names: N/A (Not applicable)
Drug: Placebo — Sodium chloride 0.9% for injection will be used as a placebo. A 1ml volume will be drawn up into a suitable sized syringe and labelled in accordance with standard practice at site. The dose will be administered as a subcutaneous injection in line with the Secukinumab/ Bimekizumab/ Ixekizumab dosing regimen. No dose adjustments are permitted.
  Other Names: N/A (Not applicable)

SUMMARY:
The investigators seek clinically actionable understanding of the mechanisms that underlie depression in the context of immune mediated inflammatory diseases (IMIDs), delivered by a focused immune intervention study examining brain circuitry using state of the art imaging in the context of exquisitely specific therapeutic immune interception in human immune disease.

Glutamate concentration in the NAcc will be positively correlated with the magnitude of the inflammatory response and will be attenuated by IL-17A inhibition. Ultimately, this will be associated with an improvement in depressive symptoms.

The strength of coupling between early and late systems will be attenuated in the context of IL-17A-driven inflammation and will be correlated with less frequent switching behaviour following negative outcomes and ultimately depressive symptoms. This coupling will be re-established following IL-17 antagonism.

Patients whose depressive symptoms benefit most from IL-17A antagonism will exhibit greatest resting-state and task-specific functional connectivity between Th-NAcc.

DETAILED DESCRIPTION:
Approximately 30-40% of patients with immune-mediated inflammatory diseases (IMIDs), such as psoriatic disease, experience depression. These symptoms negatively affect clinical outcomes, quality of life and treatment adherence. There is accumulating evidence that peripheral inflammation may contribute to the origins of depression. In particular, a) stimulation of active phase inflammation results in remitting-relapsing depressive symptoms b) abnormal neural connectivity linked to this depression is correlated with peripheral inflammation and c) biologic therapies targeting specific peripheral inflammation components (cytokines) improve depressive symptoms.

In this proposal, psoriatic disease (PsD), encompassing both psoriasis and PsA, will be our IMID exemplar. In this condition, the IL-23/IL-17 cytokine axis is central to pathogenesis, as proven by successful application of inhibitors to this pathway. Moreover, this axis has also recently been implicated in the neurobiology of depression in both preclinical and clinical studies.

The investigators aim to uncover the mechanisms that underlie depression in the context of IMIDs, delivered by a focused immune intervention study examining brain circuitry using state of the art imaging in the context of exquisitely specific therapeutic immune interception in human immune disease.

The rationale for this study is to use this specific therapeutic immune intervention to leverage mechanistic understanding of brain changes that drive depressive symptoms. Prior animal studies have clearly demonstrated the deleterious effects of proinflammatory cytokines on neural functioning. The investigators will integrate current therapy with innovative neuroimaging technologies to obtain data for the first time in humans that have hitherto only been possible in animal studies.

The intervention tools proposed herein (secukinumab, bimekizumab or Ixekizumab) are IL-17 inhibitors licensed for treatment of active PsO and PsA. Secukinumab, bimekizumab and Ixekizumab are widely used in clinical practice globally and across the UK as a first/second-line biologic disease modifying antirheumatic drug (DMARD), in line with national/international NICE (TA350, TA445, TA723, TA916, TA442, TA537) treatment recommendations. Secukinumab is given by self-administered subcutaneous injection weekly for the first five weeks of treatment and thereafter by monthly maintenance injections. Bimekizumab is given by self-administered subcutaneous injection 4 weekly, Ixekizumab is given by self -administered subcutaneous injection either 2 or 4 weekly. Typically, depressive symptoms are attenuated within weeks of therapeutic initiation. Prior study data indicate a beneficial effect of IL17 antagonism on depressive symptoms, but the mechanism of action has not yet been explored.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years < 75years
* Diagnosis of PsO or PsA, made by a dermatologist or rheumatologist.
* Selected to start secukinumab/ bimekizumab/ Ixekizumab as part of their standard clinical care by their usual dermatology team for PsO or rheumatology clinical team for PsA in line with the license for secukinumab/ bimekizumab/ Ixekizumab and NICE/SMC criteria.
* No contraindications to MRI (for example metal fragments or implantable devices not compatible with MRI. (no extra x-ray images will be obtained to check placement of metal fragments or clips insitu. Existing images may be used to check for possible contraindications)
* Satisfactory completion of standard pre-biologic safety screening (including, but not limited to, exclusion of latent TB infection according to local protocol, chest X-ray, negative HIV screen, negative Hepatitis screen antibody, negative Hepatitis B surface antigen [Hep B sAg] and negative Hepatitis B anti-core antibody [Hep B cAb])
* Recent (but not within 4 weeks prior baseline) use of intra-muscular or intra-articular steroid injections
* Women of Child-Bearing Potential (WoCBP) must be willing to use effective contraception for study duration. Further information is provided in appendix 1.
* Willing to participate and give informed consent

Exclusion Criteria:

* Inability to provide written informed consent
* Severe physical impairment (e.g., blindness, deafness, paraplegia).
* Clinically important, active infections e.g. active TB
* History of inflammatory bowel disease
* Pregnant or breast feeding
* Severe claustrophobia precluding MRI
* Contraindications to 7T MRI (metal implants in the ears, head or neck, microbladed/ tattooed eyebrows, metal fragments in the eyes)
* Confounding neurological disease including MS, Stroke, Traumatic Brain Injury
* Previous exposure to IL-17A, IL-17A/F, IL-17R inhibitors or IL-23 p19/p40 inhibitors in the last 6 months
* Hypersensitivity to any of the excipients in secukinumab/ bimekizumab/ ixekizumab.
* Any reason which, at the investigator's discretion, would make them unsuitable to take part in the study.

Ages: 18 Years to 74 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 50 participants with active PsD attending clinics in NHS Greater Glasgow and Clyde, NHS Grampian, NHS Lothian, NHS Tayside, NHS Lanarkshire, NHS Forth Valley starting IL-17 antagonism as part of their usual care by either their NHS dermatology clinical care team for psoriasis, or NHS rheumatology clinical care team for PsA, and in line with the licence and SMC/NICE guidance for these agents. The decision to prescribe anti-IL17 treatment for active PsD will be made by the patients' clinical team in advance, and independently, of the study.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Changes in glutamate concentration in the NAcc as measured by 7T MRS. | Week 0 to Week 6
  Changes in glutamate concentration in the NAcc as measured by 7T MRS, from Week 0 to Week 6 (before and after IL17 antagonism).

SECONDARY OUTCOMES:
Differences in the EEG amplitude during positive and negative response outcomes. | Week 0 to Week 6
  Changes in the EEG amplitude between the thalamic and NAcc learning systems before and after IL-17 antagonism.
Correlating fMRI signals with differences in EEG amplitude. | Week 0 to Week 6
  fMRI signals that correlate with the changing EEG amplitude, before and after IL17 antagonism.

OTHER OUTCOMES:
Changes in fatigue following IL-17 antagonism using BRAF Severity | Week 0 to Week 6
  Symptoms measured using Bristol Rheumatoid Arthritis Fatigue Severity (BRAF Severity).
Changes in fatigue following IL-17 antagonism using PROMIS-Fatigue | Week 0 to Week 6
  Symptoms measured using Patient-Reported Outcomes Measurement Information System - Fatigue (PROMIS-Fatigue).
Changes in Hyperalgesia following IL-17 antagonism using American College of Rheumatology Fibromyalgia scale. | Week 0 to Week 6
  Symptoms measured using American College of Rheumatology Fibromyalgia scale.
Changes in Pain following IL-17 antagonism using Pain-NRS. | Week 0 to Week 6
  Symptoms measured using the Numeric Rating Scale for Pain (Pain-NRS).
Changes in Pain following IL-17 antagonism using McGill Pain Questionnaire. | Week 0 to Week 6
  Symptoms measured using the McGill Pain Questionnaire.
Changes in Pain following IL-17 antagonism using Michigan Body Map Regional Pain Intensity | Week 0 to Week 6
  Symptoms measured using the Michigan Body Map Regional Pain Intensity.
Changes in Sleep Disturbance following IL-17 antagonism using PROMIS- Sleep related impairment. | Week 0 to Week 6
  Symptoms measured using the Patient-Reported Outcomes Measurement Information System - Sleep Related Impairment (PROMIS- Sleep related impairment).
Changes in Mood following IL-17 antagonism using HADS. | Week 0 to Week 6
  Symptoms measured using the Hospital Anxiety Depression Scale (HADS).
Changes in Mood following IL-17 antagonism using PROMIS-Depression. | Week 0 to Week 6
  Symptoms measured using the Patient-Reported Outcomes Measurement Information System - Depression (PROMIS-Depression).
Changes in Mood following IL-17 antagonism using PROMIS-Anxiety. | Week 0 to Week 6
  Symptoms measured using the Patient-Reported Outcomes Measurement Information System - Anxiety (PROMIS-Anxiety).
Changes in Cognition following IL-17 antagonism using Cognitive Failures Questionnaire. | Week 0 to Week 6
  Symptoms measured using the Cognitive Failures Questionnaire (CFQ).
Changes in measures of disease activity in patients with Psoriatic Arthritis before and after IL-17 antagonism using DAPSA. | Week 0 to Week 6
  Changes in measures of disease activity in patients with Psoriatic Arthritis before and after IL-17 antagonism as measured by the Disease Activity in Psoriatic Arthritis (DAPSA).
Changes in measures of disease activity in patients with Psoriatic Arthritis before and after IL-17 antagonism using PsAID-12. | Week 0 to Week 6
  Changes in measures of disease activity in patients with Psoriatic Arthritis before and after IL-17 antagonism as measured by the 12-item Psoriatic Arthritis Impact of Disease (PsAID-12).
Changes in measures of disease activity in patients with Psoriatic Arthritis or Psoriasis before and after IL-17 antagonism using PASI. | Week 0 to Week 6
  Changes in measures of disease activity in patients with Psoriatic Arthritis before and after IL-17 antagonism as measured by the Psoriasis Area and Severity Index (PASI)
Changes in measures of disease activity in patients with Psoriatic Arthritis or Psoriasis before and after IL-17 antagonism using BSA. | Week 0 to Week 6
  Changes in measures of disease activity in patients with Psoriatic Arthritis before and after IL-17 antagonism as measured by the Body Surface Area (BSA).
Changes in measures of disease activity in patients with Psoriatic Arthritis before and after IL-17 antagonism using 66/68 Joint Count. | Week 0 to Week 6
  Changes in measures of disease activity in patients with Psoriatic Arthritis before and after IL-17 antagonism as measured by the 66/68 Joint Count.
Changes in measures of disease activity in patients with Psoriatic Arthritis before and after IL-17 antagonism using DLQI. | Week 0 to Week 6
  Changes in measures of disease activity in patients with Psoriasis before and after IL-17 antagonism as measured by the Dermatology life Quality Index (DLQI).
Changes in peripheral immune biomarkers in patients before and after IL-17 antagonism. | Week 0 to Week 6
  Changes in peripheral immune biomarkers in patients before and after IL-17 antagonism.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Cavanagh, MD, PhD, Principal Investigator — University of Glasgow
Locations (1):
- Queen Elizabeth University Hospital, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Analysed by the study team at University of Glasgow.